CLINICAL TRIAL: NCT01004185
Title: A Randomized, Double-blind, Parallel-group Study to Assess the Safety and Efficacy of Asacol® (1.2 to 4.8g/Day) 400 mg Delayed-release Tablets Given Twice Daily for 26 Weeks to Children and Adolescents for the Maintenance of Remission of Ulcerative Colitis
Brief Title: Assessing the Safety/Efficacy of Asacol® Given Every 12 Hours to Children and Adolescents for the Maintenance of Remission of Ulcerative Colitis
Acronym: CAMPIII
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pediatric enrollment very slow.
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008085
Record Dates: First submitted 2009-10-27; First posted 2009-10-29 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Dose (Experimental): 2.0 - 4.8 g/day Asacol dependent on body weight
  Interventions: Drug: Asacol 400 mg
- Low Dose (Experimental): 1.2 - 2.4 g/day Asacol dependent upon body weight
  Interventions: Drug: Asacol 400 mg

INTERVENTIONS:
Drug: Asacol 400 mg — 17-33kg = 3 Asacol 400mg AM & 2 Asacol 400mg PM; 33-<54kg = 5 Asacol 400 mg AM & 4 Asacol 400mg PM; 54-<90kg = 6 Asacol 400mg AM & PM
  Other Names: mesalamine; 5-aminosalicylic acid; 5-ASA; mesalazine
  Arms: High Dose
Drug: Asacol 400 mg — 17-<33kg = 2 Asacol 400mg & 1 placebo AM, 1 Asacol 400mg & 1 placebo PM; 33-<54kg = 3 Asacol 400mg & 2 placebo AM, 2 Asacol 400mg & 2 placebo PM; 54-<90kg = 3 Asacol 400mg & 3 placebo AM & PM
  Other Names: mesalamine; 5-aminosalicylic acid; 5-ASA; mesalazine
  Arms: Low Dose

SUMMARY:
The purpose of this study is to determine whether low dose Asacol® (27 mg/kg - 71 mg/kg) and high dose Asacol® (53 mg/kg - 118 mg/kg) are safe and effective when dosed as 400 mg delayed-release tablets given twice daily for 26 weeks to children and adolescents for the maintenance of remission of ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* male or female between the ages of 5 and 17 years, inclusive, at the time of the first dose of study medication;
* have a documented history of UC that has been successfully maintained in complete remission for at least 1 month prior to study entry
* have a baseline PUCAI score < 10
* have a body weight no less than 17 kg and no more than 90 kg
* have a history of at least 1 active episode or relapse in the last 12 months
* have taken a stable maintenance dose of oral mesalamine (or equivalent oral 5-ASA dose) for at least 1 month prior to entry in the study. Stable is defined as the same dose for the last month.
* maintained complete remission, as defined, throughout the 30-day run-in phase. Note:ONLY applies to those patients who complete the 6-week treatment in complete remission from Study 2007017 and immediately roll-over to the 30-day run-in phase
* are female patients who are pre-menarchal or have a negative urine pregnancy test and, if sexually active, practice acceptable contraception (e.g., abstinence; oral, intramuscular, or implanted hormonal contraception [at least 3 months prior to enrollment]

Exclusion Criteria:

* have a history of allergy or hypersensitivity to salicylates, aminosalicylates, or any component of the Asacol tablet
* have a significant co-existing illness or other condition(s), including but not limited to cancer or significant organic or psychiatric disease on medical history or physical examination, that, in the judgment of the Investigator, contraindicate(s) administration of the study drug and/or any study procedures
* have a history or presence of any condition causing malabsorption or an effect on gastrointestinal motility or history of extensive small bowel resection (greater than one half the length of the small intestine) causing short bowel syndrome
* any "condition" causing "malabsorption" or an effect on gastrointestinal "motility"
* have current renal disease, or a screening blood urea nitrogen (BUN) or creatinine value that is > 1.5 times the upper limit of the age appropriate normal
* have a documented history of or current hepatic disease, or liver function tests (alanine transaminase [ALT], aspartate transaminase [AST], total bilirubin) that are > 2 times the upper limit of normal
* have a history of pancreatitis
* have undergone treatment with any oral, intravenous, intramuscular, or rectally administered corticosteroids (including budesonide) within 30 days prior to the Screening visit
* have undergone treatment with any rectal mesalamine therapy within 30 days prior to the screening visit
* have undergone treatment with immunomodulatory therapy including, but not limited to: rosiglitazone, 6-mercaptopurine or azathioprine, cyclosporine, or methotrexate within 90 days prior to Screening visit
* have undergone treatment with biologic therapy including, but not limited to: infliximab,adalimumab, certolizumab or other biologic treatment of ulcerative colitis within 90 days prior to Screening visit
* have undergone treatment with antibiotics (other than topical antibiotics) including metronidazole within 7 days prior to the Screening visit
* have undergone treatment with aspirin or other nonsteroidal anti-inflammatory drugs NSAIDs) within 7 days prior to the Screening visit
* have undergone treatment with any antidiarrheals and/or antispasmodics within 30 days of the Screening visit
* have a stool examination positive for Clostridium difficile (C. difficile), bacterial pathogens, or ova and parasites. Note: Because normal gut flora may vary by geography, the Medical Monitor should be consulted before excluding a patient with a stool sample that is positive for C. difficile, bacterial pathogens or ova and parasites.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Warner Chilcott
Locations (45):
- United States (24):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Loma Linda, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Park Ridge, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Portland, Maine
  - Research Site, Boston, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Southfield, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Mays Landing, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Providence, Rhode Island
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Huntington, West Virginia
- Canada (5):
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
- Croatia (2):
  - Research Site, Rijeka
  - Research Site, Zagreb
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Iași
- Russia (5):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Smolensk

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening began on 6 Oct 2009
Pre-assignment Details: There was a 30-day run-in phase for subjects continuing directly from Study 2007017.
Groups:
- High Dose: Subjects who weigh 17-<33 kg will receive 2.0 g/day Asacol. Subjects who weigh 33-<54 kg will receive 3.6 g/day Asacol. Subjects who weigh 54-<90 kg will receive 4.8 g/day Asacol.
- Low Dose: Subjects who weigh 17-<33 kg will receive 1.2 g/day Asacol. Subjects who weigh 33-<54 kg will receive 2.0 g/day Asacol. Subjects who weigh 54-<90 kg will receive 2.4 g/day Asacol.
Period: Overall Study
Arm/Group | High Dose | Low Dose
Started | 19 | 20
Completed | 10 | 11
Not Completed | 9 | 9
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Sponsor Terminated Study | 4 | 5
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Low Dose | Total
Number analyzed (Participants) | 19 | 20 | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 13.1 (2.5) | 13.2 (2.1) | 13.1 (2.3)
Age, Customized [Number; unit: participants]
  5-8 years | 1 | 0 | 1
  9-17 years | 18 | 20 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 16 | 17 | 33
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success PUCAI (Pediatric Ulcerative Colitis Activity Index), mITT/Modified Intent to Treat Population
Description: PUCAI Score (0-85, sum of scores for each): abdominal pain (0/5/10 - no pain/ignored/not ignored), rectal bleeding (0/10/20/30 - none, small amount <50% of stools, small amount most stools, large amount >50%), stool consistency (0/5/10 - formed, partially formed, completely formed), # stools/24 hrs. (0/5/10/15 - 0-2/3-5/6-8/>8), nocturnal bowel/any diarrhea causing wakening (0/10 - no/yes), activity level (0/5/10 - no limitation/occ limitation, severe restrictions). Remission <10, Mild 10-34, Moderate 35-64, Severe 65-85. Remission defined as Treatment Success.
Time Frame: Week 26
Population: MITT subjects who took at least one dose of study medication and did not have baseline stool exam positive for C. difficile, bacterial pathogens or ova/parasites.
Measure: Number; unit: percentage of participants
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 19 | 20
percentage of participants | 53.3 | 60

2. Secondary Outcome: Treatment Success PUCAI Amended Endpoint (5 Point Scale Abdominal Pain), mITT
Description: PUCAI Score (0-85, sum of scores for each) abdominal pain (0/2.5/5/7.5/10 - no pain/very mild/mild/moderate/severe), rectal bleeding (0/10/20/30 - none, small amount <50% of stools, small amount most stools, large amount >50%), stool consistency (0/5/10 - formed, partially formed, completely formed), # stools/24 hrs. (0/5/10/15 - 0-2/3-5/6-8/>8), nocturnal bowel/any diarrhea causing wakening (0/10 - no/yes), activity level (0/5/10 - no limitation/occ limitation, severe restrictions). Remission <10, Mild 10-34, Moderate 35-64, Severe 65-85. Remission is Treatment Success.
Time Frame: Week 26
Population: mITT Subjects who took at least one dose of study medication and did not have baseline stool examination positive for C. difficile, bacterial pathogens or ova/parasites.
Measure: Number; unit: percentage of participants
Arm/Group | High Dose | Low Dose
Number analyzed (Participants) | 19 | 20
percentage of participants | 60 | 60

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | High Dose | Low Dose
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/20
Other Adverse Events (participants affected / at risk) | 13/19 | 11/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (N=19) | Low Dose (N=20)
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose (N=19) | Low Dose (N=20)
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Lip Blister (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Axillary Pain (General disorders) | 1 | 0
Cyst (Gastrointestinal disorders) | 0 | 1
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 1
Cellulitis Orbital (Infections and infestations) | 1 | 1
Ear Infection (Infections and infestations) | 1 | 0
Infectious Mononucleosis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1
Viral Infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Lipase Increased (Investigations) | 1 | 1
Stool Analysis Abnormal (Investigations) | 0 | 1
Urinary Sediment Present (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Erosion (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less